CLINICAL TRIAL: NCT02022124
Title: Open Label Placebo in the Treatment of Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital de Egas Moniz (Other)
Responsible Party: Principal Investigator, Claudia Carvalho, Principal Investigator, Hospital de Egas Moniz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 88/CES-2013
Record Dates: First submitted 2013-11-21; First posted 2013-12-27 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Low Back Pain
Keywords: chronic low back pain; open-label placebo
MeSH Terms: interventions — microcrystalline cellulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- microcrystalline cellulose (open-label inert substance) (Experimental): 3-week course of non-deceptive placebo using placebo pills plus the usual regime that the patients had been prescribed at the time of intake.
  Interventions: Drug: Microcrystalline cellulose (open-label inert substance)
- Usual care treatment (No Intervention): This arm will entail a 3-week course of the stable treatment the patient is following at time of intake.

INTERVENTIONS:
Drug: Microcrystalline cellulose (open-label inert substance) — The intervention will be an inert substance, microcrystalline cellulose in a capsule. Participants will take two capsules daily.
  Arms: microcrystalline cellulose (open-label inert substance)

SUMMARY:
Patients will be randomized to receive open-label (honestly described placebo) immediately at baseline or be eligible to receive the open-label treatment three weeks after the baseline measurements. Therefore all patients will be eligible to receive open-label placebo treatment for their chronic low back pain during the course of the study.

DETAILED DESCRIPTION:
Chronic low back pain (cLBP) is a debilitating and costly condition that affects 1.2 million Portuguese with an estimated cost in the United Stated of $50 billion. Randomized controlled trials has shown that placebo interventions can dramatically reduce chronic low back pain and its associated disability. Generally, it is assumed that response to placebo requires concealment or deception, which presents a dilemma to the clinician. In clinical practice, how can patients benefit from an available, effective and potentially cost-effective intervention without being deceived? This study seeks to determine ethically acceptable open-label placebo treatment (with full informed consent) can lead to meaningful benefits. The primary study will involve 80 patients with cLBP who will be randomly assigned to a three-week course of either non-deceptive open-label placebo pills in the context of a persuasive rationale + treatment as usual or to be continued on their treatment-as-usual. Primary outcome measures will be pain intensity and symptom bothersomeness on the previous week. Additionally, the study will investigate a possible association between the genetic variation of the catechol-O-methyltransferase (COMT polymorphisms) with the hypothesized observed placebo effect on cLBP patients. Participants will be followed for 3 weeks with a mid-point (11 days) visit. Patients who receive only usual care for the first three weeks will be eligible to elect a three week course of treatment with open-label placebo after which they will be assessed. This study has been submitted and approved by the following review board: Comissão de Ética do Centro Hospitalar de Lisboa Ocidental (Lisbon West Hospitals Centre's Ethical Committee) Institutional Review Board.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years or older
* Low back pain complaints for a min. of 3 months

Exclusion Criteria:

* use of strong opioid analgesic and/or anticonvulsant medication;
* specific causes of back pain namely cancer, fractures and infections;
* complicated back problems (e.g. prior back surgery);
* conditions making treatment difficult (e.g. paralysis, psychoses);
* conditions that might confound treatment effects or interpretation of results (e.g. severe fibromyalgia, rheumatoid arthritis);
* concurrent care from other providers;
* conditions that affect safety of patient (e.g. pregnancy);
* concurrent medical legal issues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
pain intensity | previous week
  assessed by an 11-point Numeric Rating Scale (NRS)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Carvalho, PhD, Principal Investigator — ISPA - Instituto Universitario de Ciencias Psicologicas, Sociais e da Vida
Locations (1):
- Hospital de Egas Moniz, Lisbon, Portugal